CLINICAL TRIAL: NCT01756300
Title: A Prospective, Multi-Center, Non-Randomized Feasibility Study of Catheter-Based Renal Denervation to Treat Resistant Hypertension (RENABLATE- EC12-02)
Brief Title: RENABLATE Feasibility Study CS156 (EC12-02) Study of Catheter Based Renal Denervation to Treat Resistant Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RENABLATE
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Hypertension, Renal
Keywords: Essential Hypertension; Renal Denervation; Vascular Disease; Renal Catheter Ablation; Primary Hypertension
MeSH Terms: conditions — Hypertension, Renal; Essential Hypertension; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resistant Hypertension (Experimental): The catheter-based (device: Celsius® ThermoCool® RD) renal denervation will serve to treat resistant hypertension.
  Interventions: Device: Celsius® ThermoCool® RD

INTERVENTIONS:
Device: Celsius® ThermoCool® RD — The investigational device is designed to transmit radiofrequency (RF) current to the electrodes for ablation purposes, specifically for the treatment of resistant hypertension by renal denervation.
  Other Names: Multi-electrode Ablation Catheter

SUMMARY:
The RENABLATE feasibility study is a prospective, multi-center, non-randomized feasibility study to evaluate the safety and effectiveness of the investigational multi-electrode ablation catheter and integrated ablation system to treat resistant hypertension.

DETAILED DESCRIPTION:
The RENABLATE feasibility study CS156 (EC12-02) is a prospective, multi-center, non-randomized feasibility study to evaluate the safety and effectiveness of renal artery sympathetic denervation using the investigational Celsius® ThermoCool® Renal Denervation (RD) Multi-electrode Ablation Catheter and integrated ablation system to treat resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 and < 85 years old.
2. Individual has a systolic blood pressure ≥ 160 mmHg (≥ 150 mmHg for type 2 diabetics) based on an average of 3 office blood pressure readings.
3. Individual is adhering to a stable drug regimen of at least 3 different classes of anti-hypertensive medications, including a diuretic (with no changes for a minimum of 2 weeks prior to enrollment) at optimal dose and is expected to be maintained for at least 6 months.
4. Individual agrees to have all study procedures performed, and is competent and willing to provide written, informed consent to participate in this study.

Exclusion Criteria:

1. Subjects with known/diagnosed secondary hypertension.
2. Subject has 'White Coat' hypertension defined as 24 hour daytime systolic blood pressure <135 mm Hg as evaluated at Baseline visit.
3. Subject has aorto-ilio-femoral artery anatomy not suitable for treatment with the investigational Celsius® ThermoCool® RD Multi-electrode Ablation Catheter.
4. Subject has main renal arteries that are < 20 mm in length or < 4 mm in diameter.
5. Subject has multiple main renal arteries in either kidney.
6. Subject has a history of prior renal artery intervention including balloon angioplasty, stenting or surgery.
7. Subject had a previous kidney transplant or is a planned recipient of a transplant kidney or is on dialysis.
8. Subject has a past history of unilateral kidney removal or has a solitary functional kidney for any other reason.
9. Subject has an estimated glomerular filtration rate (eGFR) of < 45mL/min/1.73m2, using the MDRD formula.
10. Subject has type 1 diabetes mellitus.
11. Subject has history of Myocardial Infarction, unstable angina pectoris, or a cerebrovascular accident in the 6 months period prior to enrolment, or documented widespread atherosclerosis, intravascular thrombosis or unstable plaques.
12. Subject had a significant surgery or cardiovascular intervention in the 6 months period preceding enrollment or is planned to have such a surgery or cardiac intervention in the 6 months period post enrollment.
13. Subject has hemodynamically significant valvular heart disease for which reduction of blood pressure would be considered hazardous.
14. Subject is taking systemic steroids or chronic daily NSAIDs.
15. Subject has a known allergy to Aspirin and/or other procedural drugs or contrast agents which in the investigator's opinion excludes him/her from the study.
16. Subject has a serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study (e.g., subjects with active systemic infection, subjects with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, hemophilia, or significant anemia).
17. Women of childbearing potential with a positive pregnancy test during screening OR women who do not agree to remain on birth control until follow-up at 6 months OR lactating women.
18. Subject has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.
19. Subject is currently enrolled in another investigational drug or device trial.

Ages: 19 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2015-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrollment took approximately 11 months, began in December 2, 2012 and completed on November 4, 2013. A total of 68 subjects were consented and 35 started the renal denervation with the investigational ablation catheter.
Pre-assignment Details: After signing the inform of consent, subjects were evaluated on inclusion/exclusion criteria, anatomic eligibility, compliant with completing the subject diary. Thirty-three subjects failed and never underwent insertion of the study ablation catheter.
Groups:
- Renal Sympathetic Denervation: Subjects enrolled in this study underwent the renal sympathetic denervation procedure to treat resistant hypertension. The procedure used the investigational Celsius® ThermoCool® Renal Denervation Multi-electrode Ablation Catheter in subjects with severe resistant hypertension.
Period: Overall Study
Arm/Group | Renal Sympathetic Denervation
Started | 35 (Subjects underwent renal denervation treatment with the study catheter.)
Completed | 33 (Subjects with follow up available at 12 months)
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All treated subjects who underwent the renal sympathetic denervation procedure.
Groups:
- Renal Sympathetic Denervation: Subjects enrolled in this study underwent the renal sympathetic denervation procedure to treat resistant hypertension. The procedure used the investigational Celsius® ThermoCool® Renal Denervation Multi-electrode Ablation Catheter in subjects with resistant hypertension.
Arm/Group | Renal Sympathetic Denervation
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 23
Race/Ethnicity, Customized [Number; unit: participants]
  African Descent | 0
  Not African Descent | 35
Region of Enrollment [Number; unit: participants]
  Czech Republic | 12
  Belgium | 5
  Denmark | 1
  Australia | 15
  Italy | 2

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Major Cardiovascular and/or Renal Adverse Events Related to the Renal Denervation Procedure That Occurred Within 30 Days Post-procedure.
Description: The major adverse events include Acute myocardial infarction, Death from progressive heart failure, death from aortic or peripheral artery disease, from renal failure and sudden cardiac death, New-onset heart failure, Stroke, Aortic or lower limb, revascularization procedure, Lower limb amputation, Beginning dialysis, Hospital admission for hypertensive emergency unrelated to non-adherence or non-persistence with drugs at each follow up visit, Hospitalization for atrial fibrillation.
Time Frame: 30 days post-procedure
Population: The Safety Analysis population, which consists of all enrolled subjects who have undergone insertion of the study ablation catheter.
Measure: Number; unit: percentage of participants
Arm/Group | Renal Sympathetic Denervation
Number analyzed (Participants) | 35
percentage of participants | 0.0

2. Secondary Outcome: Subjects Experienced Any Adverse Cardiovascular and Renal Events Through 12 Months Post-procedure
Description: These adverse events include renal artery stenosis (≥60% diameter reduction confirmed by MRI or renal angiography); periprocedural renal artery dissection or perforation requiring intervention, serious arterial access site related complications requiring intervention or prolonging hospitalization; ≥25% reduction between baseline and 12 months in renal function measured by the estimated Glomerular Filtration Rate (eGFR), as well as composite of major adverse cardiovascular and/or renal events.
Time Frame: 12 months post-procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Renal Sympathetic Denervation
Number analyzed (Participants) | 35
percentage of participants | 74.3

3. Secondary Outcome: Actual and Change in Office Systolic Blood Pressure and Diastolic Blood Pressure From Baseline to 1 ,3, 6 and 12 Months Post Procedure
Description: This secondary effectiveness endpoint is defined as actual and change in office systolic blood pressure and diastolic blood pressure from baseline to 1 ,3, 6 and 12 months post procedure. Negative values represent reduction from baseline.
Time Frame: From baseline to 1 ,3, 6 and 12 months post procedure
Population: The Effectiveness analysis population, which consists of all enrolled subjects who have had technical success without major protocol deviations. Technical Success is defined to be when the investigational catheter has been successfully inserted into the femoral artery and radiofrequency (RF) energy is successfully applied in at least one artery. .
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Blood Pressures at Baseline: Office blood pressures measured at Baseline
- Blood Pressures at 1-Month Follow Up: Office blood pressures measured at one month post-procedure
- Blood Pressures at 3-Month Follow Up: Office blood pressures measured at 3-month post procedure
- Blood Pressures at 6-Month Follow Up: Office blood pressures measured at 6-month post procedure
- Blood Pressures at 12-Month Follow Up: Office blood pressures measured at 12-month post procedure
Arm/Group | Blood Pressures at Baseline | Blood Pressures at 1-Month Follow Up | Blood Pressures at 3-Month Follow Up | Blood Pressures at 6-Month Follow Up | Blood Pressures at 12-Month Follow Up
Number analyzed (Participants) | 27 | 27 | 27 | 26 | 26
mmHg
  Systolic Office Blood Pressure | 171.0 (10.4) | 161.0 (21.1) | 159.7 (21.7) | 155.4 (15.6) | 151.0 (18.7)
  Systolic Mean Change from Baseline | NA (NA) — Not applicable at Baseline for change from Baseline measures | -10.0 (21.1) | -11.3 (21.9) | -15.4 (17.6) | -19.8 (20.7)
  Diastolic Office Blood Pressure | 95.8 (16.3) | 88.3 (15.0) | 87.5 (13) | 85.0 (11.7) | 86.4 (15.7)
  Diastolic Mean Change from Baseline | NA (NA) — Not applicable at Baseline for change from Baseline measures | -7.6 (13.7) | -8.3 (12.4) | -10.7 (13.5) | -9.0 (12.9)

4. Secondary Outcome: Actual and Change in 24-hour Ambulatory Blood Pressure Monitoring (ABPM) Systolic Blood Pressure and Diastolic Blood Pressure From Baseline to 3, 6 and 12 Months Post Procedure
Description: This secondary effectiveness endpoint is defined as change in 24-hour ABPM systolic blood pressure and diastolic blood pressure from baseline to 3, 6 and 12 months post procedure. The blood pressures were measured using the 24-hour Ambulatory Blood Pressure Monitoring system. Reported values are the arithmetic mean of collected blood pressure values over 24 hours. Negative values represent reduction from baseline.
Time Frame: From baseline to 3, 6 and 12 months post procedure
Population: The Effectiveness analysis population, which consists of all enrolled subjects who have had technical success without major protocol deviations. Technical Success is defined to be when the investigational catheter has been successfully inserted into the femoral artery and RF energy is successfully applied in at least one artery. .
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Blood Pressures at Baseline: ABPM blood pressures measured at Baseline
- Blood Pressures at 3-Month Follow Up: ABPM blood pressures measured at 3-month post procedure
- Blood Pressures at 6-Month Follow Up: ABPM blood pressures measured at 6-month post procedure
- Blood Pressures at 12-Month Follow Up: ABPM blood pressures measured at 12-month post procedure
Arm/Group | Blood Pressures at Baseline | Blood Pressures at 3-Month Follow Up | Blood Pressures at 6-Month Follow Up | Blood Pressures at 12-Month Follow Up
Number analyzed (Participants) | 27 | 26 | 26 | 26
mmHg
  Systolic Office Blood Pressure | 156.0 (12.9) | 145.4 (17.2) | 142.1 (15.6) | 141.2 (15.6)
  Systolic Mean Change from Baseline | NA (NA) — Not applicable at Baseline for change from Baseline measures | -9.8 (12.7) | -13.1 (15.7) | -14.7 (14.9)
  Diastolic Office Blood Pressure | 85.8 (12.7) | 80.8 (10.8) | 78.5 (11.9) | 79.0 (11.2)
  Diastolic Mean Change from Baseline | NA (NA) — Not applicable at Baseline for change from Baseline measures | -3.9 (8.2) | -6.8 (8.0) | -7.1 (6.7)

5. Secondary Outcome: Incidence of Subjects Achieving Target Systolic Blood Pressure at 1, 3, 6, and 12 Month Post-procedure
Description: This endpoint is defined as incidence of subjects achieving target systolic blood pressure at 1, 3, 6, and 12 month post-procedure. Target systolic blood pressure is defined as less than 140 mmHg (and less than 130 mmHg for Type II Diabetics).
Time Frame: At 1, 3, 6, and 12 month post-procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Groups:
- At One Month: Subjects achieved target systolic blood pressure, i.e., less than 140 mmHg, at one month post-procedure
- At Three Month: Subjects achieved target systolic blood pressure, i.e., less than 140 mmHg, at three month post-procedure
- At Six Month: Subjects achieved target systolic blood pressure, i.e., less than 140 mmHg, at six month post-procedure
- At Twelve Month: Subjects achieved target systolic blood pressure, i.e., less than 140 mmHg, at twelve month post-procedure
Arm/Group | At One Month | At Three Month | At Six Month | At Twelve Month
Number analyzed (Participants) | 27 | 27 | 26 | 26
percentage of participants | 14.8 | 18.5 | 15.4 | 23.1

6. Secondary Outcome: Incidence of Subjects Achieving at Least 10 mmHg Systolic Blood Pressure Reduction From Baseline at 1, 3, 6, and 12 Month Post-procedure
Description: This endpoint is defined as Incidence of subjects achieving at least 10 mmHg systolic blood pressure reduction from Baseline at 1, 3, 6, and 12 month post-procedure
Time Frame: At 1, 3, 6, and 12 month post-procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Groups:
- At One Month: Subjects achieved at least 10 mmHg systolic blood pressure reduction from Baseline at one month post-procedure
- At Three Month: Subjects achieved at least 10 mmHg systolic blood pressure reduction from Baseline at three month post-procedure
- At Six Month: Subjects achieved at least 10 mmHg systolic blood pressure reduction from Baseline at six month post-procedure
- AT Twelve Month: Subjects achieved at least 10 mmHg systolic blood pressure reduction from Baseline at Twelve month post-procedure
Arm/Group | At One Month | At Three Month | At Six Month | AT Twelve Month
Number analyzed (Participants) | 27 | 27 | 26 | 26
percentage of participants | 48.1 | 48.1 | 61.5 | 76.9

ADVERSE EVENTS:
Time Frame: Twelve months post procedure
Arm/Group | Renal Sympathetic Denervation
Serious Adverse Events (participants affected / at risk) | 7/35
Other Adverse Events (participants affected / at risk) | 23/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Sympathetic Denervation (N=35)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 2 (2)
Sudden death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Sympathetic Denervation (N=35)
Albumin urine high (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3)
Breathlessness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Flu-like illness (General disorders) | 1 (1)
Function kidney decreased (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertension worsened (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 3 (3)
Incision site bleeding (Injury, poisoning and procedural complications) | 1 (1)
Incision site hematoma (Injury, poisoning and procedural complications) | 3 (3)
Inflammation (General disorders) | 1 (1)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Middle ear infection (Infections and infestations) | 1 (1)
Numbness (Nervous system disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Painful knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1)
Raised blood pressure (Investigations) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 3 (3)
Renal function test (Investigations) | 1 (1)
Serum potassium decreased (Investigations) | 1 (1)
Serum sodium decreased (Investigations) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spasm of artery (Vascular disorders) | 4 (4)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Swelling arm (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Urethral irritation (Renal and urinary disorders) | 1 (1)
Vertebral artery stenosis (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.